CLINICAL TRIAL: NCT05481827
Title: ORACLE: A Long-term Follow-up Study to Evaluate the Safety of GT005 in Participants With Geographic Atrophy Secondary to Age-related Macular Degeneration Treated in a Gyroscope-sponsored Antecedent Study
Acronym: ORACLE
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Gyroscope Therapeutics Limited (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GT-ORACLE; 2020-003987-22 (EudraCT Number); CPPY988A12203B (Other: Novartis)
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Age Related Macular Degeneration (AMD)
Keywords: Geographic Atrophy; Retinal disease; Retinal degeneration; Macular atrophy; Dry age-related macular degeneration; Macular degeneration; age-related macular degeneration (ARMD); retina damage; dry macular degeneration; AMD
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy; Retinal Diseases; Retinal Degeneration; Anetoderma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GT005 (Experimental): GT005 is a gene therapy for GA and is a recombinant adeno-associated viral serotype 2 (AAV2) vector encoding for human complement factor I. GT005 was administered to all participants in an antecedent study prior to enrollment in ORACLE and GT005 is not administered in the ORACLE study
  Interventions: Genetic: GT005

INTERVENTIONS:
Genetic: GT005 — GT005 is a gene therapy for GA and is a recombinant adeno-associated viral serotype 2 (AAV2) vector encoding for human complement factor I. GT005 was administered to all participants in an antecedent study prior to enrollment in ORACLE and GT005 is not administered in the ORACLE study.

SUMMARY:
The purpose of this study is to evaluate the long-term safety of GT005 in participants with Geographic Atrophy (GA) secondary to AMD who have been treated in an antecedent study.

DETAILED DESCRIPTION:
This is a prospective, multi-centre, long-term, follow-up study for participants who have previously received GT005 in one of the antecedent clinical studies which were prematurely terminated GT005-01 (FOCUS), GT005-02 (EXPLORE) or GT005-03 (HORIZON). Participants from GT005-01 (FOCUS) study with only 1 last study visit to be conducted (Week 240) will remain in the study to complete their last visit. No investigational product will be administered within this study, and participants will be invited to enter ORACLE upon their completion or termination of the antecedent interventional study (whichever is soonest). This study will consist of up to three study visits prior to Week 96, and up to five study visits thereafter, for an overall period of 5-years post-GT005 administration.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent
2. Received GT005 in an antecedent study, GT005-01 (FOCUS, NCT03846193), GT005-02 (EXPLORE, NCT04437368) and GT005-03 (HORIZON, NCT04566445)
3. Willing to attend study visits and complete the study procedures.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2028-06-02 (Estimated); Study Completion 2028-06-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular and systemic adverse events (AEs) | up to Week 260
  An AE is the development of an undesirable medical condition or the deterioration of a preexisting medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the IMP.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (21):
  - Retina Consultants San Diego - Poway, Poway, California
  - Southwest Retina Research Center, Durango, Colorado
  - Vitreo Retinal Associates Pa - the Millennium Center Location, Gainesville, Florida
  - Rand Eye Institute, Inc. (Rei), Pompano Beach, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - University Retina and Macula Associates, P.C. - Lemont Office, Lemont, Illinois
  - Midwest Eye Institute Northside, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - The Retina Care Center, Llc - Baltimore Location, Baltimore, Maryland
  - Ophthalmic Consultants of Boston (OCB), Boston, Massachusetts
  - Pepose Vision Institute, P.C - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Columbia University Medical Center, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Sterling Vision - Oregon Retina, Llp, Eugene, Oregon
  - Mid Atlantic Retina - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Retina Consultants of Austin, Austin, Texas
  - Texas Retina Associates (Tra) - Dallas Main, Dallas, Texas
  - Retina Consultants of Texas (Retina Consultants of Houston) - Texas Medical Center, Houston, Texas
  - Retinal Consultants of San Antonio (Rcsa) - Medical Center, San Antonio, Texas
- The University of Melbourne - The Centre for Eye Research Australia (CERA), Melbourne E., Victoria, Australia
- France (2):
  - CHU Dijon - Hopital Mitterrand, Dijon
  - CHU de Nantes - Hôtel-Dieu, Nantes
- Germany (2):
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
  - Universitaetsklinikum Tuebingen, Tübingen
- Spain (3):
  - Instituto de microcirugía ocular, Barcelona
  - Clinica Baviera, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
- United Kingdom (2):
  - The Retina Clinic London, London
  - South Tyneside and Sunderland Nhs Foundation Trust - Sunderland Eye Infirmary, Sunderland